CLINICAL TRIAL: NCT07000929
Title: The Use of Videonystagmography With Caloric Testing as an Instrumental Diagnostic Method for Vestibular Migraine
Brief Title: Videonystagmography and Vestibular Migraine
Status: Recruiting | Type: Observational
Sponsor: Dr. med. Lukas Becker (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Lukas Becker, Principal Investigator, Universitätsklinikum Essen
Organization: Universitätsklinikum Essen (Other)
Other Study IDs: VM_LB_DHL
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Migraine Disorders; Vertigo
Keywords: Vestibular migraine; Vertigo; Migraine; Dizziness
MeSH Terms: conditions — Migraine Disorders; Vertigo; Dizziness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vestibular migraine confirmed: Patients who received a diagnosis of vestibular migraine.
  Interventions: Diagnostic Test: Videonystagmography
- Episodic or chronic migraine, without vestibular migraine: Patients who received a diagnosis of episodic or chronic migraine without vestibular migraine.
  Interventions: Diagnostic Test: Videonystagmography
- Healthy participants: Patients who not received a diagnosis of episodic or chronic migraine nor vestibular migraine.
  Interventions: Diagnostic Test: Videonystagmography

INTERVENTIONS:
Diagnostic Test: Videonystagmography — In the regular examination of patients with vertigo, videonystagmography with thermal testing (caloric) is already an established and necessary examination procedure that is used to diagnose many different vertigo disorders.

SUMMARY:
In the study, the investigators would like to examine whether there is a difference between patients with vestibular migraine, patients with episodic or chronic migraine and healthy subjects in the examination of videonystagmography, which has been used for many years to differentiate and diagnose vertigo disorders. Accordingly, videonystagmography could also be discussed as an important diagnostic instrument for the diagnosis of the still young disease vestibular migraine.

DETAILED DESCRIPTION:
Vestibular migraine is a young disorder that is caught between headache experts and vertigo experts. In 2012, the International Bárány Society for Neurootology and the International Headache Society were able to agree on a uniform definition and terminology for "vestibular migraine" in a jointly formulated consensus paper. A distinction is currently made between "definite" and "probable" vestibular migraine on the basis of the applicable diagnostic criteria. The diagnostic criteria are based on a study from 2001 with 75 patients and a follow-up period of 8 years, in which the diagnosis was confirmed in 84% of cases. At present the diagnostic criterion still requires the exclusion of another possible vestibular or ICHD diagnosis. Vestibular migraine is reported in the literature as the most common cause of spontaneous episodic vertigo attacks in adults and children. A manifestation is basically possible at any age. Despite the frequency of vestibular migraine and the sometimes pronounced level of suffering, the publication density is low and the diagnosis is mainly based on the patient medical history and clinical neurological examination. No specific instrumental diagnostic method or specific biomarkers that confirm or even prove the diagnosis are known. Larger studies with the intention of improving the diagnosis and thus achieving the expected reduction in the postulated high number of unreported cases have not yet been carried out. In the regular examination of patients with vertigo, videonystagmography with caloric testing is already an established and necessary examination procedure that is used to diagnose many different vertigo disorders. In the investigations, patients with confirmed vestibular migraine often show a vestibular hyperexcitability or increased caloric reaction not previously described in the literature. The investigators would like to verify this with this study. The investigators therefore developed the hypothesis of a possible correlation between a certain nystagmus frequency and/or certain speed of the slow phase of the nystagmus and the presence of a vestibular migraine. Comparisons with patients with headache migraine without accompanying vertigo symptoms and with a healthy control group should be carried out to test the hypothesis. First, all patients at the Dizziness Center at University Hospital Essen with diagnosed vestibular migraine without other conditions, except episodic or chronic migraine, were analyzed in the first quarter of 2023. This was followed by the inclusion of patients with episodic or chronic migraine and no vestibular migraine, standardized by age and gender, as well as the inclusion of a healthy control group without migraine headache and without vestibular migraine. Following that the collected data will be analyzed in particular the videonystagmography with caloric testing and the comparison of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: The diagnosis of vestibular migraine is confirmed.
* Group 2: The diagnosis of episodic or chronic migraine is confirmed. There is no coexisting vestibular migraine.
* Group 3: healthy subjects without vestibular migraine and episodic or chronic migraine

Exclusion Criteria:

* Simultaneous presence of another confirmed vertigo disorder
* A previous hearing loss
* Simultaneous presence of a chronic disease that affects the sense of balance
* Taking medication with a central effect that affects the sense of balance
* An existing eardrum defect or a blocked ear canal due to earwax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of patients was recruited from the dizziness center of the University Hospital Essen. The patients with migraine were recruited partly from the headache center and partly via advertising. The healthy subjects were recruited through advertising.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
mean comparison nystagmus frequency | Mean of nystagmus frequency at study enrollment, Baseline
  Comparison of the mean between the group of patients with vestibular migraine and the patients and healthy participants in the mean nystagmus frequency within 30 seconds
mean comparison GLP (speed of the slow phase) of nystagmus in °/s or sum of °/s | Mean of nystagmus GLP at study enrollment, Baseline
  Comparison of the mean between the group of patients with vestibular migraine and the patients and healthy participants in the mean GLP of nystagmus in °/s or sum of °/s
Comparison head impulse test (vHIT) | result of head impulse test at study enrollment, Baseline
  Comparison of the mean between the group of patients with vestibular migraine and the patients and healthy participants in the qualitativ analysis of the head impulse test

CONTACTS AND LOCATIONS:
Overall Officials: Dagny Holle-Lee, Prof. Dr. med., Study Director — Klinik für Neurologie, Universitätsklinikum Essen
Locations (1):
- Westdeutsches Kopfschmerz und Schwindelzentrum der Klinik für Neurologie des Universitätklinikums Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Disclosure of personal hospital data was not agreed in the ethics vote. The patient was informed with the indication that the data would not be passed on.

REFERENCES:
- [Background] Rocha MF, Sacks B, Al-Lamki A, Koohi N, Kaski D. Acute vestibular migraine: a ghost diagnosis in patients with acute vertigo. J Neurol. 2023 Dec;270(12):6155-6158. doi: 10.1007/s00415-023-11930-9. Epub 2023 Aug 19. No abstract available. PMID 37597072
- [Background] Muelleman T, Shew M, Subbarayan R, Shum A, Sykes K, Staecker H, Lin J. Epidemiology of Dizzy Patient Population in a Neurotology Clinic and Predictors of Peripheral Etiology. Otol Neurotol. 2017 Jul;38(6):870-875. doi: 10.1097/MAO.0000000000001429. PMID 28498271
- [Background] Lempert T, Olesen J, Furman J, Waterston J, Seemungal B, Carey J, Bisdorff A, Versino M, Evers S, Newman-Toker D. Vestibular migraine: diagnostic criteria. J Vestib Res. 2012;22(4):167-72. doi: 10.3233/VES-2012-0453. PMID 23142830